CLINICAL TRIAL: NCT00370929
Title: Treatment of Epilepsy by Meditation and Cultivation of Emotional Balance
Brief Title: A Study of Meditation as a Treatment for Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, John Stern, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSPC-06-03-001
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Meditation (Experimental)
  Interventions: Behavioral: Meditation

INTERVENTIONS:
Behavioral: Meditation

SUMMARY:
Epileptic seizures may occur at times of stress and commonly increase life stress. This study will evaluate whether meditation improves seizure control and quality of life for individuals with uncontrolled epilepsy.

DETAILED DESCRIPTION:
Individuals who have uncontrolled epilepsy commonly experience disability, depression, anxiety and injuries from seizures. For such individuals, ideal treatments should improve quality of life through control of seizures and improved emotional state. Meditation with cultivation of emotional balance is known to improve emotional state and may also benefit seizure control in some individuals. In this study, individuals with uncontrolled epilepsy will receive detailed training in meditation to determine whether the training leads to improvements in seizure control and various measures of emotion and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 6 or more seizures per month
* ability to participate in meditation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Seizure frequency | 20 weeks
Quality of Life | 20 weeks

SECONDARY OUTCOMES:
Mood | 20 weeks
Affect | 20 weeks
Anxiety | 20 weeks
Sleep quality | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Stern, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Geffen School of Medicine at UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No